CLINICAL TRIAL: NCT06095921
Title: The Effect of Self-Management Programme Performed Via Telerehabilitation on Occupational Performance and Satisfaction of Individuals With Systemic Sclerosis
Brief Title: The Effect of a Self-Management Program on Individuals With Scleroderma
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Emirhan Karakuş (Other)
Responsible Party: Sponsor-Investigator, Emirhan Karakuş, Director, Hacettepe University
Organization: Hacettepe University (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: ERG-EMIRHAN-001
Record Dates: First submitted 2023-10-15; First posted 2023-10-23 (Actual); Last update posted 2023-10-23 (Actual); Status verified 2023-10

CONDITIONS: Scleroderma; Systemic Sclerosis
MeSH Terms: conditions — Scleroderma, Diffuse; Scleroderma, Systemic

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Our employee's statistical analysis was conducted by a biostatistician unrelated to her work.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Self Management Intervention Program (Experimental): That program was created by sending 40-minute videos 1 day a week for 8 weeks. The programme was developed both according to the achievements of previous self-management studies and according to the occupations that individuals with SSc have difficulty with.
  Interventions: Behavioral: Self Management Intervention Program
- Statistical Analysis (No Intervention): One week after the program, the biostatistician evaluated the results.

INTERVENTIONS:
Behavioral: Self Management Intervention Program — SSc, the course of the disease, symptoms and coping strategies, medications and treatment methods? The importance of exercise for individuals with SSc, and how to create an action plan for an exercise? were discussed. What are fatigue and its symptoms? How can we protect our articular-energy and how should a quality rest be? What is pain and what are coping approaches? What is the pain-related area of influence? What are body image problems, how to use problem solving approach and what is its importance? What is Stress? What is mindfulness? What are mindfulness exercises? What are the ways to cope with stress? What are the daily life occupations and how can we facilitate them? How can we solve problems in difficult occupations? How to create an occupation plan to facilitate daily occupations? What are oral stretching exercises and how to do them? What are the factors affecting sleep? What is advocacy and why is it important? Answers to these questions were sought.
  Arms: Self Management Intervention Program

SUMMARY:
Introduction: Individuals with systemic sclerosis (SSc) have problems with perceived occupational performance and satisfaction in daily life activities due to many symptoms caused by the disease.

Purpose: This study will plan to examine the effect of a self-management program for individuals with SSc on perceived occupational performance and satisfaction.

Materials and Methods : Twenty-nine individuals with SSC, 28 females and 1 male will participate in the study. Perceived occupational performance and satisfaction levels before and after the program will evaluate with the Canadian Ocupational Performance Measure (COPM). The training programme will design according to the activities of COPM, the needs of the patients, and the literature. The programme consists of 8 sessions for 8 weeks, 1 day a week for 45 minutes.

DETAILED DESCRIPTION:
In this study, 36 individuals, diagnosed with scleroderma by a rheumatologist at Gazi University, were included. In the study approved by the Gazi University Clinical Research Ethics Committee (21.09.2020, Decree No: 635) and planned by the Declaration of Helsinki, consent forms were sent to all participants to confirm that they were volunteers. Demographic information of the individuals was obtained. The Canadian Occupational Performance Measure (COPM) was used to identify occupational problems and to implement a person-centered program. This information was obtained by submitting online forms. The videos were prepared by a team of physiotherapists, occupational therapists, and rheumatology doctors. The program manager was an occupational therapist. 29 people completed the 8-week program, which included 40-50 minute videos and assignments (keeping a pain diary, creating an exercise routine, etc.). At the end of the program, individuals were reminded of the difficult occupations again so that the Canadian Occupational Performance Measure could be re-scored. Initially, the open-ended question "In which ways did the program contribute to you?" was asked. Individuals were evaluated in the first and last week of the program and the results were compared. These evaluations and interventions were made during the Covid-19 pandemic.

ELIGIBILITY:
Inclusion Criteria:

Clinical diagnosis of Scleroderma's Disease, being in remission period for 6 months, being between the ages of 18-65, knowing how to use technological devices.

Exclusion criteria:

Neurological disease, continuing a different study or rehabilitation programme, having COVID-19 infection, exacerbation the disease in the last 6 months.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2020-07-15 (Actual); Primary Completion 2020-10-15 (Actual); Study Completion 2021-01-15 (Actual)

PRIMARY OUTCOMES:
Canadian Occupational Performance Measurement (COPM) | One week before the rehabilitation program is implemented.
  COPM was developed in 1990. The scale determines the daily life occupations experienced by individuals in the areas of self-care, productivity and leisure time. It grades the occupational performance and satisfaction points of these determined occupations according to the Likert scale between 1-10. A minimum of one and a maximum of 5 occupations could be written, resulted in a total performance and satisfaction point. The average performance and satisfaction points were divided by the number of readings. The highest point that can be obtained from the scale is 10 and the lowest point is 1. The Turkish cultural adaptation, validity and reliability study of the scale was conducted by Torpil in 2017 in individuals with multiple sclerosis and the test-retest reliability of the Turkish version was found to be 0.98.
Canadian Occupational Performance Measurement (COPM) | One week after the rehabilitation program ended.
  COPM was developed in 1990. The scale determines the daily life occupations experienced by individuals in the areas of self-care, productivity and leisure time. It grades the occupational performance and satisfaction points of these determined occupations according to the Likert scale between 1-10. A minimum of one and a maximum of 5 occupations could be written, resulted in a total performance and satisfaction point. The average performance and satisfaction points were divided by the number of readings. The highest point that can be obtained from the scale is 10 and the lowest point is 1. The Turkish cultural adaptation, validity and reliability study of the scale was conducted by Torpil in 2017 in individuals with multiple sclerosis and the test-retest reliability of the Turkish version was found to be 0.98.

CONTACTS AND LOCATIONS:
Locations (1):
- Hacettepe University, Çankaya, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No